CLINICAL TRIAL: NCT02172755
Title: Single-dose and Steady-state Pharmacokinetics of BIA 2-093 and Its Metabolites in Healthy Elderly Subjects Compared With Those in Healthy Young Subjects
Brief Title: Single-dose and Steady-state Pharmacokinetics of BIA 2-093 and Its Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-105
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Epilepsy
Keywords: Eslicarbazepine acetate; BIA 2-093
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly subjects (Experimental): 14 Elderly subjects aged 65 years or more; During the whole study, subjects were to receive a single 600 mg dose of BIA 2-093 (Phase A) followed by 600 mg BIA 2-093 once daily for 8 days in Phase B. Phase B was to begun 96 hours post-Phase A dose.
  Interventions: Drug: BIA 2-093
- Young subjects (Experimental): 16 young subjects aged between 18 and 40 years During the whole study, subjects were to receive a single 600 mg dose of BIA 2-093 (Phase A) followed by 600 mg BIA 2-093 once daily for 8 days in Phase B. Phase B was to begun 96 hours post-Phase A dose.
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093 — During the whole study, subjects were to receive a single 600 mg dose of BIA 2-093 (Phase A) followed by 600 mg BIA 2-093 once daily for 8 days in Phase B. Phase B was to begun 96 hours post-Phase A dose.
  Other Names: Eslicarbazepine acetate

SUMMARY:
The purpose of this study is to determine the effects of age on the pharmacokinetic profile of BIA 2-093 and its active metabolites.

DETAILED DESCRIPTION:
This was a single-centre, open-label, parallel group, non-randomised study with a single-dose phase (Phase A) followed by a multiple-dose phase (Phase B), in 12 healthy elderly and 12 healthy young subjects. During the whole study, subjects were to receive a single 600 mg dose of BIA 2-093 (Phase A) followed by 600 mg BIA 2-093 once daily for 8 days in Phase B. Phase B was to begun 96 hours post-Phase A dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 40 years, inclusive OR male or female subjects aged 65 years or more.
* If young, subjects who were within 15% of ideal body weight OR, if elderly, subjects who were within 20% of ideal body weight according to the Metropolitan Life Insurance Table.
* Subjects who were healthy as determined by pre-study medical history, physical examination, neurological examination, and 12-lead ECG.
* Subjects who had clinical laboratory tests acceptable to the Investigator.
* Subjects who were negative for HBsAg, HCVAb and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for alcohol and drugs of abuse at screening.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or menopause or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine.
* (If female and with less than 40 years old) She had a negative pregnancy test at screening.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used drugs within 2 weeks of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of their first admission to this study.
* Subjects who had previously received BIA 2-093.
* Subjects who had donated and/or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding
* (If female) She was of childbearing potential and she did not use an authorised effective contraceptive method.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-06; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Scope International Life Sciences AG,, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elderly Subjects | Young Subjects
Started | 14 | 16
Completed | 12 | 12
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly Subjects | Young Subjects | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 15 | 15
  >=65 years | 14 | 0 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration (Cmax)
Description: Single-dose period: Day 1 at pre-dose, and ½, 1, 1½, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours post-dose.
  Multiple-dose period: from Day 5 to Day 11 inclusive, early in the morning, before the daily dose (for trough levels).
  Day 12: pre-dose, and ½, 1, 1½, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post-last dose.
  BIA 2-194, BIA 2-195, and oxcarbazepine are metabolites of BIA 2-093
Time Frame: Day 1 at pre-dose, and ½, 1, 1½, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours post-dose From Day 5 to Day 11 inclusive, before the daily dose (for trough levels). On Day 12, pre-dose, and ½, 1, 1½, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours p
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Elderly Subjects | Young Subjects
Number analyzed (Participants) | 12 | 12
ng/mL
  Single dose (BIA 2-194) | 9469 (2284) | 9867 (1714)
  Multiple dose (BIA 2-194) | 15067 (2126) | 17309 (3430)
  Single dose (BIA 2-195) | 209 (72.1) | 192 (31.5)
  Multiple dose (BIA 2-195) | 531 (190) | 461 (132)
  Single dose (oxcarbazepine) | 76.3 (29.5) | 77.3 (15.6)
  Multiple dose (oxcarbazepine) | 135 (36.6) | 150 (36.6)

2. Secondary Outcome: Tmax - Time of Maximum Observed Concentration
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Elderly Subjects | Young Subjects
Number analyzed (Participants) | 12 | 12
hours
  Single dose (BIA 2-194) | 2.96 (1.25) | 3.00 (1.81)
  Multiple dose (BIA 2-194) | 2.04 (0.916) | 2.04 (1.57)
  Single dose (BIA 2-195) | 13.6 (5.43) | 11.3 (6.57)
  Multiple dose (BIA 2-195) | 7.29 (4.18) | 7.58 (2.68)
  Single dose (oxcarbazepine) | 5.41 (3.29) | 5.41 (2.96)
  Multiple dose (oxcarbazepine) | 2.67 (1.54) | 2.67 (1.48)

3. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve to Last Measurable Time Point
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Elderly Subjects | Young Subjects
Number analyzed (Participants) | 12 | 12
ng.h/mL
  Single dose (BIA 2-194) | 190521 (69082) | 174713 (37062)
  Multiple dose (BIA 2-194) | 288364 (40878) | 290630 (68649)
  Single dose (BIA 2-195) | 5738 (3675) | 3361 (1295)
  Multiple dose (BIA 2-195) | 15911 (4852) | 12782 (3722)
  Single dose (oxcarbazepine) | 1014 (965) | 577 (246)
  Multiple dose (oxcarbazepine) | 1508 (725) | 1490 (495)

ADVERSE EVENTS:
Arm/Group | Elderly Subjects | Young Subjects
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/16
Other Adverse Events (participants affected / at risk) | 11/14 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderly Subjects (N=14) | Young Subjects (N=16)
cardiovascular collapse (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elderly Subjects (N=14) | Young Subjects (N=15)
Tiredness (General disorders) | 8 | 8
Headache (Nervous system disorders) | 5 | 4
Dizziness (Nervous system disorders) | 0 | 3
Concentration impaired (Nervous system disorders) | 1 | 1
Drowsiness (Nervous system disorders) | 0 | 1
Head pressure (Nervous system disorders) | 0 | 1
Vision blurred (Nervous system disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea with vomiting (Gastrointestinal disorders) | 0 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 1
Exanthema (Skin and subcutaneous tissue disorders) | 1 | 1
Decrease activity (Psychiatric disorders) | 1 | 0
Sinus pressure (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other